CLINICAL TRIAL: NCT04873180
Title: A Retrospective Study
Brief Title: Significance of Immunohistochemical Expression of Survivin in Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-21-04-28
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Survivin; Immnuohistochemistry
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue sections from cases of renal tumors will be preserved in formalin fixed, parraffin embedded blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sectioning and staining of renal neoplasms after nephrectomy operation — nephrectomy operations will be done to patients diagnosed as having renel tumors

SUMMARY:
detection of Survivin expression in renal cell carcinoma and correlate this expression to tumor grade and stage.

DETAILED DESCRIPTION:
renal cell carcinoma is the third most prevalent malignant tumor of the genitourinary system. deregulation of apoptosis is involved in carcinogenesis by abnormally prolonged cell survival, facilitating accumulations of multiple mutations and augment resistance to immune-surveillance. Survivin is a member of inhibitor of Apoptosis Protein family (IAPs). it play a role in cell cycle regulation by inhibiting apiptosis. Survivin is over-expressed in many human neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* patients suffer from renal cell carcinomas

Exclusion Criteria:

* patients received pre-operative chemotherapy or radiotherapy. patients with insufficient clinical data.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms and signs of renal neoplasms admitted to Sohag University hospital and underwent nephrectomy operations. excisional specimens sent to pathology Lab will be sectioned and stained by H&E. only cases of renal cell carcinoma will be included in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
expression of survivin in neoplastic and adjacent normal renal tissues | april, 2021
  Survivin is highly expressed in neoplastic renal tissues compared to normal ones by immunohistochemical measures..

CONTACTS AND LOCATIONS:
Overall Officials: Maisa H Mohammed, MD, Principal Investigator — a lecturer of pathology, Sohag faculty of medicine
Locations (1):
- Maisa Hashem Mohammed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided